CLINICAL TRIAL: NCT04361565
Title: Prevalence and Clinical Evolution of Olfactory and Taste Disorders in Patients Infected by SARS-CoV-2
Brief Title: Frequency and Clinical Evolution of Olfactory and Taste Disorders in COVID-19 Patients
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 20odontocovid01
Record Dates: First submitted 2020-04-22; First posted 2020-04-24 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: COVID-19 by SARS-CoV-2 Infection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Individuals diagnosed for COVID-19

SUMMARY:
A novel coronavirus SARS-CoV-2 HAS arose in 2019 in Wuhan, China. Beside the classical semiology of this infection, numerous patients described olfactory and teste disorders. These symptoms are not described in this coronavirus, neurotropism of coronaviridae has been documented before. The aim of the study is to evaluate prevalence of anosmia and dysgeusia (olfactory and taste disorders) in coronavirus diagnosed patients and compare with different clinical conditions. The second endpoint is to evaluate the duration of these symptoms in order to better understand the semiology of this infection.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 diagnosed

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals that responded to a online form
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2020-03-20 (Actual); Primary Completion 2020-04-10 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Anosmia | 45 days
  Prevalence for anosmia in the COVID-19 + patients
Ageusia | 45 days
  Prevalence for ageusia in the COVID-19 + patients
Duration of the loss of anosmia ageusia | 45 days
  Duration measured in days

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nice, Nice, France